CLINICAL TRIAL: NCT01773304
Title: Acute Effects of Dairy and Meat Proteins on Bone Metabolism and Metabolic Profile in Urine and Plasma in Overweight Adults
Brief Title: Acute Effects of Dairy and Meat Proteins on Bone Metabolism and Metabolic Profile
Acronym: MEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Agriculture and Food Council (Other)
Responsible Party: Principal Investigator, AAstrup, Dr Med Sci, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: M210
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Obesity; Bone Metabolism
Keywords: Obesity; Adults; Bone metabolism; Metabolic profile; Dairy protein; Meat protein
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meal rich in dairy protein (Experimental)
  Interventions: Other: Dietary meal intervention
- Meal rich in meat protein (Experimental)
  Interventions: Other: Dietary meal intervention

INTERVENTIONS:
Other: Dietary meal intervention — Test meals with different protein types (dairy versus meat)

SUMMARY:
The purpose of this randomized, controlled, cross over single meal study is to investigate the metabolic effects of a breakfast rich in dairy proteins and to determine biomarkers for their intake. The results from this project will increase our knowledge about nutritional value of dairy proteins, which is necessary to decide whether dairy products can be recommended for prevention of weight related bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 18 and 50 years
* BMI 25-40

Exclusion Criteria:

* Physical activity more than 10 hours weekly
* Smoking
* Diagnosed osteoporosis in at least one parent
* Dietary supplements and vitamin pills (during the study and 2 months before the start)
* Vegetarians and vegans
* Lactose intolerant
* Women who are pregnant, breastfeeding or post-menstrual
* Regular intake of medication
* Chronic diseases (including osteoporosis, cancer, diabetes, cardiovascular disease and mental disorders)
* Participation in other clinical trials that could affect the test results
* Donation of blod within 3 months before intervention start
* Hypersensitivity to paraaminobenzoic acid (PABA)
* Not able to comply with the procedures established by the Protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
serum C-terminal carboxy-terminal collagen crosslinks (CTX) | at 0, 30, 60, 120, 180 and 240 min at both visits
urine C-terminal carboxy-terminal collagen | baseline 24-h urine samples and 24-h urine samples after the meal test at both visits
serum osteocalcin (sOC) | at 0, 30, 60, 120, 180 and 240 min at both visits
serum tartrate-resistant acid phosphatase (s-TRAP) | at 0, 30, 60, 120, 180 and 240 min at both visits
urine deoxypyridinoline crosslink (uDPD) | baseline 24-h urine samples and 24-h urine samples after the meal test at both visits
plasma metabolites for metabolomics analyses | at 0, 30, 60, 120, 180 and 240 min at both visits
urine metabolites for metabolomics analyses | baseline 24-h urine samples, 24-h urine samples after the meal test, urine samples at 2-h and 4-h after the meal test and urine samples from 4-h to 24-h, all at both visits

SECONDARY OUTCOMES:
serum insulin-growth factor-1 (IGF-1) | at 0, 30, 60, 120, 180 and 240 min at both visits
serum insulin-growth factor binding-protein-3 (IGFBP-3) | at 0, 30, 60, 120, 180 and 240 min at both visits
serum insulin | at 0, 30, 60, 120, 180 and 240 min at both visits
serum glucose | at 0, 30, 60, 120, 180 and 240 min at both visits
serum glukagon-like peptide-1 (GLP-1) | at 0, 30, 60, 120, 180 and 240 min at both visits
urinary PABA | baseline 24-h urine samples and 24-h urine samples after the meal test at both visits
urinary creatinin | baseline 24-h urine samples and 24-h urine samples after the meal test at both visits
urinary biobank | baseline 24-h urine samples and 24-h urine samples after the meal test at both visits
plasma biobank | at 0, 30, 60, 90, 120, 180 and 240 min at both visits

OTHER OUTCOMES:
weight | at baseline at both visits
height | at baseline at the first visit

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Copenhagen, Frederiksberg C, Denmark